CLINICAL TRIAL: NCT02498938
Title: Evaluation of SERPINA1 Gene Polymorphisms in COPD as a Risk Factor for Periodontitis
Brief Title: The Association of SERPINA1 Gene Disturbance in Patients With Lung and Gum Disorders
Acronym: SA1PLG
Status: Completed | Type: Observational
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr.Sneha Agarwal, P.G student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: D149206031
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Generalized Chronic Periodontitis
Keywords: Pulmonary disease,chronic obstructive,; generalized chronic periodontitis; SERPINA1 gene polymorphism
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — alpha 1-Antitrypsin; HIV Protease Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 2ml of blood sample from each subject will be collected in EDTA containing vials and kept at -20 degrees until DNA extraction. the genomic DNA will be isolated and Z/S polumorphism in SERPINA1 gene will be identified by PCR followed by restriction digestion pattern by Alu 1 restriction enzyme.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SERPINA1 gene in COPD and periodontitis: patients aged between 30-70 yrs with COPD (satisfying Gold's criteria) and chronic periodontitis (>4mm pocket probing depth)
  Interventions: Genetic: SERPINA1 gene

INTERVENTIONS:
Genetic: SERPINA1 gene — 2ml blood sample collected from patients to extract DNA for assessment of SERPINA1 gene polymorphism
  Other Names: serine peptidase inhibitor; proteinase inhibitor

SUMMARY:
Chronic obstructive pulmonary disease and periodontitis are chronic inflammatory diseases. The study aims to determine if the genetic polymorphism of SERPINA1 gene in patients with COPD serve as a risk factor for developing periodontitis.

DETAILED DESCRIPTION:
periodontitis is a polymicrobial inflammatory disease caused by various modifiable and non-modifiable risk factors. the non-modifiable risk factors include genetic polymorphisms like the gene coding for alpha-1-antitrypsinase

COPD is a chronic inflammatory disease characterized by deterioration of lung function due to loss of elasticity of the lungs.

SERPINA1 gene product has a protective role on the connective tissue components of both lungs and gums.

Hence, this study tries to determine if the gene polymorphism in COPD serves as a risk factor for developing periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 30-70yrs diagnosed with COPD and chronic periodontitis who are willing to participate in the study.

Exclusion Criteria:

* Pateints with other systemic disorders
* patients not willing to participate in the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients,both male and female aged between 30-70yrs with COPD nd chronic periodontitis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
SERPINA1 gene polymorphism | 9 months
  of blood samples and running samples by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sneha Agarwal, PG(perio), Principal Investigator — Panineeya Mahavidyalaya institute of dental sciences and research centre
Locations (1):
- Dr. Sneha Agarwal PG(periodontics), Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott DA, von Ahsen N, Palmer RM, Wilson RF. Analysis of two common alpha 1-antitrypsin deficiency alleles (PI*Z and PI*S) in subjects with periodontitis. J Clin Periodontol. 2002 Dec;29(12):1118-21. doi: 10.1034/j.1600-051x.2002.291212.x. PMID 12492914
- [Background] Travis J, Pike R, Imamura T, Potempa J. The role of proteolytic enzymes in the development of pulmonary emphysema and periodontal disease. Am J Respir Crit Care Med. 1994 Dec;150(6 Pt 2):S143-6. doi: 10.1164/ajrccm/150.6_Pt_2.S143. PMID 7952650